CLINICAL TRIAL: NCT06839950
Title: Sensory Profile and Early Clinical Signs of Calm Room Users
Acronym: EVAL-APAISE
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Esquirol (Other)
Responsible Party: Principal Investigator, Aude Paquet, Psychomotor Therapist, Doctor in Psychology, Centre Hospitalier Esquirol
Other Study IDs: EVAL-APAISE; 2023-A00580-45 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2025-02-12; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Psychotic Disorders; Personality Disorders; Mood Disorders
Keywords: Calm room; Psychotic Disorders; Sensory Profile; Mood Disorders; Personality Disorders
MeSH Terms: conditions — Psychotic Disorders; Personality Disorders; Mood Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

INTERVENTIONS:
Other: Calm room — The calm room combines the effects of music, light, and videos designed with natural atmospheres. Four themes are offered in the calm room: Comfort, Optimism, Freshness, and Lullaby. These themes feature nature videos, combining relaxing images with calm musical ambiance. The lighting can be adjusted by the user, who can choose from a varied color palette. The available lights have a low glare level, and the light intensity can also be adjusted by the user.
  They can be used by patients any time they want and for as long as they want.
  Other Names: Sensory room; Comfort room

SUMMARY:
This descriptive study aims primarily to characterize the sensory profile of patients in a closed psychiatric hospital unit who use a calming room.

The main questions it aims to answer are :

* Could sensory information processing disorders be the cause of distress and tension in these patients?
* Could users of the calming room present extreme sensory processing profiles, characterized by either hypersensitivity or hyposensitivity ?

Participants will answer a survey to determine their the sensory profile. Participants can already use the calming room as part of their regular medical care and they will answer surveys before and after each use.

ELIGIBILITY:
Inclusion Criteria:

* Gender and Age: Male or female, aged 18 to 65
* Hospitalization: Admitted to the closed hospitalization unit for less than 10 days
* Social security: Affiliated or beneficiary of a social security system
* Consent: Free, informed, and written consent, signed by the participant and/or their legal representative (for participants under protection measures) and the investigator (at the latest on the day of inclusion and before any research-related examination).

Exclusion Criteria:

* Inability to understand information related to the study
* Proven sensory disability
* Dementia
* Pregnancy
* Lack of social protection
* Previous Participation in this research protocol (in the case of a new hospitalization)
* Expression abilities incompatible with completing the AASP Scale (e.g., french language comprehension issues, mute individuals, patients in restraint and/or therapeutic isolation)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be enrolled from the Deniker unit in the Esquirol Hospital Center of Limoges, France.
  This study may involve a vulnerable population. In psychiatric settings, calming rooms are typically installed in closed units that admit crisis patients. These individuals may be hospitalized involuntarily or be under protective measures. Since the study focuses on individuals who are able to use such devices within the participating unit, they can be considered vulnerable.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2027-12-19 (Estimated); Study Completion 2028-05-19 (Estimated)

PRIMARY OUTCOMES:
Scores of Sensory Sensitivity from the Adolescent/Adult Sensory Profile (Brown and Dunn, 2002) for users of the calming room and non-users of the calming room | At enrollment
  The sensory profile scores will be obtained through the Adolescent/Adult Sensory Profile (AASP) scale during an individual interview following the participant inclusion. The following Sensory Sensitivity sub-score will be collected. The minimum and maximum values are from 15 to 75. A high score indicate a high sensory sensitivity.

SECONDARY OUTCOMES:
Scores of the Low Registration from the Adolescent/Adult Sensory Profile (Brown and Dunn, 2002) for users of the calming room and non-users of the calming room | At enrollment
  The sensory profile scores will be obtained through the Adolescent/Adult Sensory Profile (AASP) scale during an individual interview following the participant inclusion. The following Low Registration sub-score will be collected. The minimum and maximum values are from 15 to 75. A high score indicate a high Low Registration.
Scores of the Sensation Seeking from the Adolescent/Adult Sensory Profile (Brown and Dunn, 2002) for users of the calming room and non-users of the calming room | At enrollment
  The sensory profile scores will be obtained through the Adolescent/Adult Sensory Profile (AASP) scale during an individual interview following the participant inclusion. The following Sensation Seeking sub-score will be collected. The minimum and maximum values are from 15 to 75. A high score indicate a high Sensation Seeking.
Scores of the Sensation Avoiding from the Adolescent/Adult Sensory Profile (Brown and Dunn, 2002) for users of the calming room and non-users of the calming room | At enrollment
  The sensory profile scores will be obtained through the Adolescent/Adult Sensory Profile (AASP) scale during an individual interview following the participant inclusion. The following Sensation Avoiding sub-score will be collected. The minimum and maximum values are from 15 to 75. A high score indicate a high Sensation Avoiding.
Comparison of Adolescent/Adult Sensory Profile score between the user and non-user of the calming room | From enrollment to the end of observation at 2 weeks
  * Adolescent/Adult Sensory Profile scores (Sensory Sensitivity / Low Registration / Sensation Seeking / Sensory Avoidance) among calming room user
  * Adolescent/Adult Sensory Profile scores (Sensory Sensitivity / Low Registration / Sensation Seeking / Sensory Avoidance) among calming room non-user
Anxiety for users or non-user of the calming room | From enrollment to the end of observation at 2 weeks
  Anxiety is assessed from the Hamilton Anxiety Rating Scale for users and non-users of the calming room.
  The overall score ranges from 0 to 60. The generally accepted threshold for significant anxiety is 20.
Frequency of use of the calming room | From enrollment to the end of observation at 2 weeks
  - Frequency of Calming Room Use during the 14-Day Participation Period: Total number of uses of the room / time (hours)
Initiative for the use of the calming room | From enrollment to the end of observation at 2 weeks
  Modes of use of the calming room among patients who use this room.
  Qualitative measure is used for initiative :
  Patient initiative or team initiative
Reason for resquesting of the calming room | From enrollment to the end of observation at 2 weeks
  Modes of use of the calming room among patients who use this room.
  Qualitative measure is used for reason for resquesting use of the calming room :
  Anxiety / Sadness / Fatigue / Physical Tension / Seeking Well-being
Autonomy for the use of the calming room | From enrollment to the end of observation at 2 weeks
  Modes of use of the calming room among patients who use this room.
  Qualitative measure is used for autonomy for the use of the calming room :
  Presence of caregiver / Partial autonomy (one-off intervention by a caregiver) / Total autonomy (nocaregiver intervention during the use)
User frenquecy of the calming room | From enrollment to the end of observation at 2 weeks
  Number of uses of the calming room during the hospitalization
Description of anxiety leading to the use of the calming room among patients who use this room. | From enrollment to the the end of observation at 2 weeks
  Description of early clinical signs leading to the use of the calming room among patients who use this room.
  Visual Analog Score for anxiety
Description of well-being leading to the use of the calming room among patients who use this room. | From enrollment to the the end of observation at 2 weeks
  Description of early clinical signs leading to the use of the calming room among patients who use this room.
  - Visual Analog Score for well-being
Description of physical tension leading to the use of the calming room among patients who use this room. | From enrollment to the the end of observation at 2 weeks
  Description of early clinical signs leading to the use of the calming room among patients who use this room.
  - Visual Analog Score for physical tension

CONTACTS AND LOCATIONS:
Locations (1):
- Esquirol Hsopital Center, Limoges, Nouvelle-Aquitaine, France

IPD SHARING:
Plan to Share IPD: No